CLINICAL TRIAL: NCT05032053
Title: Antithrombotic Drug Use in Patients With Ischemic Stroke and Microbleeds
Acronym: AIM-2
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Ankang Central Hospital (Other); Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJLL-KY20212114
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; microbleeds; Proteomics; antithrombotic drug
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Antithrombotic drugs — The purpose of our study is to observe the effect of various antithrombotic drugs on the prognosis of ischemic stroke patients with cerebral microbleeds.

SUMMARY:
To observe the effect of different antithrombotic drugs on the prognosis of ischemic stroke patients with cerebral microbleeds. And further combined with proteomic methods to explore serological markers that can be used to accurately predict the prognosis of such patients.

DETAILED DESCRIPTION:
Cerebral microbleeds (CMBs) are caused by microvascular lesions in the brain, which is a subclinical deposition of hemosiderin after the damage of microvascular. Antithrombotic drug are widely used in the secondary prevention of patients with ischemic stroke. Studies have shown that antithrombotic drug can increase the incidence of intracranial hemorrhage in ischemic stroke patients with cerebral microbleeds. For such patients, how to carry out effective and safe antithrombotic therapy is still unclear.

We will study from two aspects: 1) We designed a cohort registration study to observe the prognosis and progress of CMBs in ischemic stroke patients one year after using various antithrombotic drugs. 2) Data independent acquisition quantitative proteomics (DIA quantitative proteomics) will be used to screen serum protein markers that may affect the prognosis of ischemic stroke patients with CMBs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed clinically as ischemic stroke;
2. Age ≥ 40 years;
3. Onset time ≤ 3 months;
4. Informed consent was signed.

Exclusion Criteria:

1. Patients with symptomatic intracranial hemorrhage;
2. bleeding lesion > 10 mm was found on SWI;
3. Vascular malformations, tumors, abscesses or other major non ischemic brain diseases were present;
4. There are contraindications for antithrombotic drugs use;
5. Serious systemic diseases;
6. Refusal to sign informed consent or poor compliance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population we observed are hospitalized patients with new cerebral infarction and met the inclusion criteria(without exclusion criteria). The method of consecutive participant sampling is used to collect the included population.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Increase of cerebral microbleeds | 1 year after onset
  How many cerebral microbleeds increased after 1 year of antithrombotic drugs treatment. The number of microbleeds will be detected by MR-SWI.

SECONDARY OUTCOMES:
Stroke recurrence rate | 1 year after onset
  recurrence rate of ischemic stroke
The incidence of cerebral hemorrhage | 1 year after onset

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, Ph.D, Study Director — Department of Neurology, Xijing Hospital, Fourth Military Medical University
Locations (16):
- China (16):
  - Ankang Central Hospital, Ankang, Shaanxi
  - 3201 Hospital, Hanzhong, Shaanxi
  - Department of Neurology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - Yan'an University Affiliated Hospital, Ya'an, Shaanxi
  - Yulin No.2 Hospital, Yunlin, Shaanxi
  - Xi'AN GAOXIN Hospital, Xi'an, Shannxi
  - Hanzhong People's Hospital, Hanzhong
  - 986 Hospital, Xi'an
  - Gaoling District Hospital, Xi'an
  - Gem Flower Xi'an Changqing Staff Hospital, Xi'an
  - Tangdu Hospital, Xi'an
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
  - No.215 Hospital of Shaanxi nuclear industry, Xianyang
  - The First People's Hospital of Xianyang, Xianyang
  - Xian Yang Central Hospital, Xianyang
  - Yan'an People's Hospital, Yan’an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson D, Ambler G, Shakeshaft C, Brown MM, Charidimou A, Al-Shahi Salman R, Lip GYH, Cohen H, Banerjee G, Houlden H, White MJ, Yousry TA, Harkness K, Flossmann E, Smyth N, Shaw LJ, Warburton E, Muir KW, Jager HR, Werring DJ; CROMIS-2 collaborators. Cerebral microbleeds and intracranial haemorrhage risk in patients anticoagulated for atrial fibrillation after acute ischaemic stroke or transient ischaemic attack (CROMIS-2): a multicentre observational cohort study. Lancet Neurol. 2018 Jun;17(6):539-547. doi: 10.1016/S1474-4422(18)30145-5. Epub 2018 May 16. PMID 29778365
- [Background] Shoamanesh A, Hart RG, Connolly SJ, Kasner SE, Smith EE, Marti-Fabregas J, Liu YY, Uchiyama S, Mikulik R, Veltkamp R, O'Donnell MJ, Ntaios G, Muir KW, Field TS, Santo GC, Olavarria V, Mundl H, Lutsep H, Berkowitz SD, Sharma M. Microbleeds and the Effect of Anticoagulation in Patients With Embolic Stroke of Undetermined Source: An Exploratory Analysis of the NAVIGATE ESUS Randomized Clinical Trial. JAMA Neurol. 2021 Jan 1;78(1):11-20. doi: 10.1001/jamaneurol.2020.3836. PMID 33074284
- [Background] Cordonnier C, Al-Shahi Salman R, Wardlaw J. Spontaneous brain microbleeds: systematic review, subgroup analyses and standards for study design and reporting. Brain. 2007 Aug;130(Pt 8):1988-2003. doi: 10.1093/brain/awl387. Epub 2007 Feb 24. PMID 17322562
- [Background] Nandigam RN, Viswanathan A, Delgado P, Skehan ME, Smith EE, Rosand J, Greenberg SM, Dickerson BC. MR imaging detection of cerebral microbleeds: effect of susceptibility-weighted imaging, section thickness, and field strength. AJNR Am J Neuroradiol. 2009 Feb;30(2):338-43. doi: 10.3174/ajnr.A1355. Epub 2008 Nov 11. PMID 19001544
- [Background] Vernooij MW, Haag MD, van der Lugt A, Hofman A, Krestin GP, Stricker BH, Breteler MM. Use of antithrombotic drugs and the presence of cerebral microbleeds: the Rotterdam Scan Study. Arch Neurol. 2009 Jun;66(6):714-20. doi: 10.1001/archneurol.2009.42. Epub 2009 Apr 13. PMID 19364926
- [Background] Liu S, Li C. Antiplatelet Drug Use and Cerebral Microbleeds: A Meta-analysis of Published Studies. J Stroke Cerebrovasc Dis. 2015 Oct;24(10):2236-44. doi: 10.1016/j.jstrokecerebrovasdis.2015.05.022. Epub 2015 Aug 10. PMID 26272868
- [Background] Lau KK, Lovelock CE, Li L, Simoni M, Gutnikov S, Kuker W, Mak HKF, Rothwell PM. Antiplatelet Treatment After Transient Ischemic Attack and Ischemic Stroke in Patients With Cerebral Microbleeds in 2 Large Cohorts and an Updated Systematic Review. Stroke. 2018 Jun;49(6):1434-1442. doi: 10.1161/STROKEAHA.117.020104. Epub 2018 May 10. PMID 29748422
- [Background] Cheng Y, Wang Y, Song Q, Qiu K, Liu M. Use of anticoagulant therapy and cerebral microbleeds: a systematic review and meta-analysis. J Neurol. 2021 May;268(5):1666-1679. doi: 10.1007/s00415-019-09572-x. Epub 2019 Oct 15. PMID 31616992
- [Background] Charidimou A, Boulouis G, Shams S, Calvet D, Shoamanesh A; International META-MICROBLEEDS Initiative. Intracerebral haemorrhage risk in microbleed-positive ischaemic stroke patients with atrial fibrillation: Preliminary meta-analysis of cohorts and anticoagulation decision schema. J Neurol Sci. 2017 Jul 15;378:102-109. doi: 10.1016/j.jns.2017.04.042. Epub 2017 Apr 28. PMID 28566143
- [Background] MRI predicts intracranial hemorrhage in patients who receive long-term oral anticoagulation. Neurology. 2019 Sep 3;93(10):465. doi: 10.1212/WNL.0000000000007920. No abstract available. PMID 31477619
- [Background] Kimura K, Aoki J, Shibazaki K, Saji N, Uemura J, Sakamoto Y. New appearance of extraischemic microbleeds on T2*-weighted magnetic resonance imaging 24 hours after tissue-type plasminogen activator administration. Stroke. 2013 Oct;44(10):2776-81. doi: 10.1161/STROKEAHA.113.001778. Epub 2013 Jul 25. PMID 23887835
- [Background] Shoamanesh A, Yan S, Charidimou A. New Cerebral Microbleeds and Mechanism of Post-Thrombolysis Remote Intracerebral Hemorrhage: "Red Meets White" Revisited. Front Neurol. 2015 Sep 15;6:203. doi: 10.3389/fneur.2015.00203. eCollection 2015. No abstract available. PMID 26441822
- [Background] Klarenbeek P, van Oostenbrugge RJ, Rouhl RP, Knottnerus IL, Staals J. Higher ambulatory blood pressure relates to new cerebral microbleeds: 2-year follow-up study in lacunar stroke patients. Stroke. 2013 Apr;44(4):978-83. doi: 10.1161/STROKEAHA.111.676619. Epub 2013 Feb 28. PMID 23449261
- [Background] Gregoire SM, Brown MM, Kallis C, Jager HR, Yousry TA, Werring DJ. MRI detection of new microbleeds in patients with ischemic stroke: five-year cohort follow-up study. Stroke. 2010 Jan;41(1):184-6. doi: 10.1161/STROKEAHA.109.568469. Epub 2009 Nov 5. PMID 19892991